CLINICAL TRIAL: NCT03548987
Title: Effect and Safety of Semaglutide 2.4 mg Once-weekly in Subjects With Overweight or Obesity Who Have Reached Target Dose During run-in Period
Brief Title: Research Study Investigating How Well Semaglutide Works in People Suffering From Overweight or Obesity
Acronym: STEP 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4376; U1111-1201-0898 (Other: World Health Organization (WHO)); 2017-003473-34 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Run-in Period: Participants will receive semaglutide at an escalating doses (0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg) for 20 weeks (week 0 to week 20). The dose will be escalated to next level every 4 weeks.
  Maintenance period: Participants will be randomized to receive semaglutide injection for 48 weeks (from week 20 to week 68).
  The trial product will be administered as an adjunct to a reduced-calorie diet and increased physical activity during the trial period.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Run-in Period: Participants will receive semaglutide at an escalating doses (0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg) for 20 weeks (week 0 to week 20). The dose will be escalated to next level every 4 weeks.
  Maintenance period: Participants will be randomized to receive semaglutide placebo injection for 48 weeks (from week 20 to week 68).
  The trial product will be administered as an adjunct to a reduced-calorie diet and increased physical activity during the trial period.
  Interventions: Drug: Semaglutide; Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous (under the skin) injection of semaglutide once-weekly.
Drug: Placebo — Subcutaneous (under the skin) injection of semaglutide placebo once-weekly.
  Arms: Placebo

SUMMARY:
This study will look at the change in participant's body weight from the start to the end of the study. This is to compare the effect on body weight in people taking semaglutide (a new medicine) and people taking "dummy" medicine. In addition to taking the medicine, the participant will have talks with study staff about healthy food choices, how to be more physically active and what a participant can do to lose weight.

The participant will get semaglutide for the first 20 weeks. Then the participant will get either semaglutide or "dummy" medicine - which treatment the participant gets after the 20 weeks is decided by chance. The participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The study will last for about 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Body mass index greater than or equal to 30 kg/sqm or greater than or equal to 27 kg/sqm with the presence of at least one of the following weight related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Haemoglobin A1c greater than or equal to 48 mmol/mol (6.5%) as measured by central laboratory at screening
* A self-reported change in body weight more than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (59):
- United States (25):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Alpharetta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Elkridge, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Wenatchee, Washington
- Denmark (2):
  - Novo Nordisk Investigational Site, Frederiksberg C
  - Novo Nordisk Investigational Site, Køge
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Netherlands (2):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Arnhem
- Portugal (5):
  - Novo Nordisk Investigational Site, Braga
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Porto
  - Novo Nordisk Investigational Site, Vila Nova de Gaia
- South Africa (4):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
- Spain (4):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Seville
- Sweden (3):
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Uppsala
- Switzerland (5):
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Olten
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Zollikerberg
  - Novo Nordisk Investigational Site, Zurich
- Ukraine (3):
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Odesa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Background] Kushner RF, Calanna S, Davies M, Dicker D, Garvey WT, Goldman B, Lingvay I, Thomsen M, Wadden TA, Wharton S, Wilding JPH, Rubino D. Semaglutide 2.4 mg for the Treatment of Obesity: Key Elements of the STEP Trials 1 to 5. Obesity (Silver Spring). 2020 Jun;28(6):1050-1061. doi: 10.1002/oby.22794. PMID 32441473
- [Result] Rubino D, Abrahamsson N, Davies M, Hesse D, Greenway FL, Jensen C, Lingvay I, Mosenzon O, Rosenstock J, Rubio MA, Rudofsky G, Tadayon S, Wadden TA, Dicker D; STEP 4 Investigators. Effect of Continued Weekly Subcutaneous Semaglutide vs Placebo on Weight Loss Maintenance in Adults With Overweight or Obesity: The STEP 4 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1414-1425. doi: 10.1001/jama.2021.3224. PMID 33755728
- [Derived] Wilkinson L, Holst-Hansen T, Laursen PN, Rinnov AR, Batterham RL, Garvey WT. Effect of semaglutide 2.4 mg once weekly on 10-year type 2 diabetes risk in adults with overweight or obesity. Obesity (Silver Spring). 2023 Sep;31(9):2249-2259. doi: 10.1002/oby.23842. PMID 37605636
- [Derived] Kosiborod MN, Bhatta M, Davies M, Deanfield JE, Garvey WT, Khalid U, Kushner R, Rubino DM, Zeuthen N, Verma S. Semaglutide improves cardiometabolic risk factors in adults with overweight or obesity: STEP 1 and 4 exploratory analyses. Diabetes Obes Metab. 2023 Feb;25(2):468-478. doi: 10.1111/dom.14890. Epub 2022 Oct 28. PMID 36200477
- [Derived] Perreault L, Davies M, Frias JP, Laursen PN, Lingvay I, Machineni S, Varbo A, Wilding JPH, Wallenstein SOR, le Roux CW. Changes in Glucose Metabolism and Glycemic Status With Once-Weekly Subcutaneous Semaglutide 2.4 mg Among Participants With Prediabetes in the STEP Program. Diabetes Care. 2022 Oct 1;45(10):2396-2405. doi: 10.2337/dc21-1785. PMID 35724304
- [Derived] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 73 sites in Denmark (2), Israel (6), Netherlands (3), Portugal (6), South Africa (6), Spain (7), Sweden (4), Switzerland (6), Ukraine (5) and United States (28).
Pre-assignment Details: The trial included 20-week run-in period and 48-week maintenance period. During the run-in period, participant started with a semaglutide dose of 0.25 mg and the dose was increased every fourth week until the target dose, 2.4 mg was reached. Out of 902 participants, 803 have completed the run-in period. Thus, these were randomised in 2:1 ratio either to receive semaglutide 2.4 mg or placebo. The treatment is an adjunct to reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide 2.4 mg: Participants were to receive once-weekly subcutaneous (s.c) injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL in 20 week run-in period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. The participants with target dose reached were randomised in 2:1 at week 20, to receive once weekly semaglutide s.c 2.4 mg until week 68.
- Placebo: Participants were to receive once-weekly s.c injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL in 20 week run-in period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. The participants with target dose reached were randomised in 2:1 at week 20, to receive once weekly placebo until week 68.
Period: Run-in Period (Week 0 to Week 20)
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 902 | 0
Safety Analysis Set (SAS) | 902 | 0
Completed | 803 | 0
Not Completed | 99 | 0
Not completed — Other | 9 | 0
Not completed — Lost to Follow-up | 8 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Safety concern as judged by investigator | 2 | 0
Not completed — Run-in failure | 19 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 48 | 0
Period: Maintenance Period (Week 20 to Week 68)
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 535 | 268
Full Analysis Set (FAS) | 535 | 268
Completed | 504 | 237
Not Completed | 31 | 31
Not completed — other | 12 | 23
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 13 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 535 | 268 | 803
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47 (12) | 46 (12) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429 | 205 | 634
  Male | 106 | 63 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 21 | 63
  Not Hispanic or Latino | 493 | 247 | 740
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 35 | 104
  White | 446 | 226 | 672
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomisation to Week 68 in Body Weight (%)
Description: Change in body weight from baseline (week 20) to week 68 is presented. The endpoint was evaluated based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75). On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Randomisation (week 20) to week 68
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Percentage point
  In-trial | -8.3 (8.1) | 6.5 (7.7)
  On-treatment: number analyzed (Participants) | 495 | 234
  On-treatment | -8.8 (7.8) | 6.1 (7.7)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -14.75, 95% CI 2-sided [-16.00 to -13.50]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Other; p < 0.0001, MMRM (mixed model repeated measurement); Treatment difference = -15.33, 95% CI 2-sided [-16.52 to -14.13]

2. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 20) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 518 | 248
Centimeter (cm) | -6.9 (7.5) | 3.2 (7.0)

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from week 20 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 518 | 248
Millimeters of mercury (mmHg) | 0 (14) | 5 (13)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from week 20 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 518 | 248
mmHg | 0 (9) | 1 (9)

5. Secondary Outcome: Change in Physical Functioning Score (Short Form 36 [SF-36])
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary and mental component summary). The 0-100 scale scores from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. Change from week 20 in the domain scores and component summary scores were evaluated at week 68. A positive change score indicates an improvement since baseline. These endpoints were evaluated based on the data from in-trial observation period which is the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 515 | 245
Scores on a scale
  Change in physical functioning score (SF-36) | 1.0 (3.8) | -1.2 (4.5)
  Change in SF-36 role-physical score | 0.3 (5.0) | -0.9 (5.3)
  Change in SF-36 bodily pain score | 0.5 (7.0) | -1.5 (7.7)
  Change in SF-36 general health score | 0.3 (5.2) | -1.8 (5.8)
  Change in SF-36 vitality score | 1.1 (7.1) | -2.1 (7.6)
  Change in SF-36 social functioning score | 0.1 (6.2) | -1.8 (6.9)
  Change in SF-36 mental health score | 0.2 (6.2) | -2.2 (7.6)
  Change in SF-36 physical component summary | 0.8 (4.9) | -0.9 (5.6)
  Change in SF-36 mental component summary | 0.0 (6.2) | -2.4 (8.5)
  Change in SF-36 role-emotional score | 0.0 (5.5) | -2.2 (7.0)

6. Secondary Outcome: Change in Body Weight [Kilogram (Kg)]
Description: Change in body weight from week 20 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomisation (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Kg | -7.5 (7.6) | 5.7 (6.7)

7. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from week 20 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/sqm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Kilogram per square meter (kg/sqm) | -2.7 (2.7) | 2.0 (2.4)

8. Secondary Outcome: Change in Haemoglobin A1c (HbA1c) [%]
Description: Change in HbA1c from week 20 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 515 | 246
Percentage point of HbA1c | -0.2 (0.3) | 0.1 (0.2)

9. Secondary Outcome: Change in HbA1c [Millimoles Per Mole (mmol/Mol)]
Description: as for outcome 8
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 515 | 246
mmol/mol | -1.7 (2.8) | 1.2 (2.7)

10. Secondary Outcome: Change in Fasting Plasma Glucose [Milligrams Per Deciliter (mg/dL)]
Description: Change in fasting plasma glucose from week 20 to week 68 is presented.The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 511 | 242
mg/dL | -1.1 (8.6) | 7.6 (10.0)

11. Secondary Outcome: Change in Fasting Plasma Glucose [Millimoles Per Litre (mmol/L)]
Description: as for outcome 10
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 511 | 242
mmol/L | -0.1 (0.5) | 0.4 (0.6)

12. Secondary Outcome: Change in Fasting Serum Insulin
Description: Change in fasting serum insulin from baseline (week 20) to week 68 [measured as milli-international units per milliliter (mIU/mL)] is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 498 | 240
Ratio of fasting serum insulin | 0.81 (60.9) | 1.03 (64.6)

13. Secondary Outcome: Change in Total Cholesterol
Description: Change in fasting total cholesterol from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 517 | 245
Ratio of fasting total cholesterol | 1.05 (13.5) | 1.11 (14.4)

14. Secondary Outcome: Change in High-density Lipoproteins (HDL)
Description: Change in fasting HDL from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 515 | 245
Ratio of fasting HDL cholesterol | 1.18 (13.2) | 1.18 (16.3)

15. Secondary Outcome: Change in Low-density Lipoproteins (LDL)
Description: Change in fasting LDL from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline.The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 517 | 245
Ratio of fasting LDL cholesterol | 1.01 (19.8) | 1.07 (21.3)

16. Secondary Outcome: Change in Very Low-density Lipoproteins (VLDL)
Description: Change in fasting VLDL from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting VLDL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 517 | 245
Ratio of fasting VLDL | 0.94 (33.6) | 1.12 (39.0)

17. Secondary Outcome: Change in Free Fatty Acids
Description: Change in fasting free fatty acids from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting free fatty acids
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 498 | 240
Ratio of fasting free fatty acids | 0.78 (79.4) | 0.89 (73.1)

18. Secondary Outcome: Change in Triglycerides
Description: Change in fasting triglycerides from baseline (week 20) to week 68 (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomization (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 517 | 245
Ratio of fasting triglycerides | 0.94 (33.9) | 1.12 (39.4)

19. Secondary Outcome: Subjects Who Achieve (Yes/no): Responder Definition Value for SF-36 Physical Functioning Score
Description: The number of participants achieving at least a 4.3-point increase in SF-36 physical functioning score from baseline (week 20) to week 68 is presented. In the reported data, 'Yes' infers number of participants who have achieved 4.3 points of increase of the score and 'No' infers number of participants who have not achieved 4.3 points of increase of the score. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomisation (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 515 | 245
Participants
  Yes | 58 | 11
  No | 457 | 234

20. Secondary Outcome: Subjects Who Gain Weight (Yes/no)
Description: The number of participants with weight gain from the start of the randomised period (week 20) to week 68 is presented. In the reported data, 'Yes' infers number of participants who have gained weight and 'No' infers number of participants who have not gained weight. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Randomisation (week 20) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Participants
  Yes | 79 | 206
  No | 441 | 44

21. Secondary Outcome: Change in Body Weight
Description: The body weight change (%) from week 0 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Run-in (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Percentage point | -17.7 (9.8) | -5.4 (7.3)

22. Secondary Outcome: Subjects Who Achieve (Yes/no): Body Weight Reduction < 0%
Description: The number of participants who achieved less than (<) 0% weight loss from week 0 to week 68 is presented. In the reported data, 'Yes' infers number of participants who have achieved <0% weight loss whereas 'No' infers number of participants who have not achieved <0% weight loss.The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Run-in (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Participants
  Yes | 22 | 51
  No | 498 | 199

23. Secondary Outcome: Subjects Who Achieve (Yes/no): Body Weight Reduction ≥ 5%
Description: The number of participants who achieved greater than or equal to (≥) 5% weight loss from week 0 to week 68 is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 5% weight loss whereas 'No' infers number of participants who have not achieved ≥ 5% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Run-in (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Participants
  Yes | 461 | 119
  No | 59 | 131

24. Secondary Outcome: Subjects Who Achieve (Yes/no): Body Weight Reduction ≥ 10%
Description: The number of participants who achieved ≥ 10% weight loss from week 0 to week 68 is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 10% weight loss whereas 'No' infers number of participants who have not achieved ≥ 10% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Run-in (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Participants
  Yes | 411 | 51
  No | 109 | 199

25. Secondary Outcome: Subjects Who Achieve (Yes/no): Body Weight Reduction ≥ 15%
Description: The number of participants who achieved ≥ 15% weight loss from week 0 to week 68 is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 15% weight loss whereas 'No' infers number of participants who have not achieved ≥ 15% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of run-in (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Run-in (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 520 | 250
Participants
  Yes | 331 | 23
  No | 189 | 227

26. Secondary Outcome: Number of Treatment-emergent Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event that had onset date (or increase in severity) on or after the first day of exposure to treatment (week 0-20 run-in period). The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week 0) to randomisation (week 20)
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 902 | 0
Events | 3775 |

27. Secondary Outcome: Number of Treatment-emergent AEs
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to treatment (week 20-75). The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Randomisation (week 20) to week 75
Population: SAS included all participants who received at least one dose of trial product. Only randomised subjects in the safety analysis set contribute.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Events | 1885 | 779

28. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. The SAEs occurred during run-in period from week 0 to week 20 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week 0) to randomisation (week 20)
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 902 | 0
Events | 23 |

29. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: as for outcome 28
Time Frame: Randomisation (week 20) to week 75
Population: as for outcome 27
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Events | 51 | 19

30. Secondary Outcome: Change in Pulse
Description: Change in pulse rate from week 0 week to week 20 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week 0) to randomisation (week 20)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
beats per minute (bpm) | 5 (9) | 5 (9)

31. Secondary Outcome: Change in Pulse
Description: Change in pulse from week 20 and 68 is presented. The endpoint was evaluated based on the data from on-treatment observation period.On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Randomisation (week 20) to week 68
Population: SAS included all participants who received at least one dose of trial product. Only randomised subjects in the safety analysis set contribute. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 495 | 234
bpm | -2 (9) | -5 (10)

32. Secondary Outcome: Change in Amylase
Description: Change in amylase (measured as units per liter [U/L]) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week) 0 to randomization (week 20)
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Ratio of amylase | 1.06 (18.7) | 1.02 (26.2)

33. Secondary Outcome: Change in Amylase
Description: Change in amylase (measured as U/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Randomisation (week 20) to week 68
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 494 | 233
Ratio of amylase | 1.06 (19.9) | 1.00 (24.9)

34. Secondary Outcome: Change in Lipase
Description: Change in lipase (measured as U/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week 0) to randomization (week 20)
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Ratio of lipase | 1.44 (40.2) | 1.39 (53.5)

35. Secondary Outcome: Change in Lipase
Description: as for outcome 34
Time Frame: Randomisation (week 20) to week 68
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 494 | 233
ratio of lipase | 0.94 (37.8) | 0.68 (51.7)

36. Secondary Outcome: Change in Calcitonin
Description: Change in calcitonin (measured as nanogram per liter (ng/L)]) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Run-in (week 0) to randomization (week 20)
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 535 | 268
Ratio of Calcitonin | 0.98 (28.4) | 0.96 (28.1)

37. Secondary Outcome: Change in Calcitonin
Description: Change in calcitonin (measured as ng/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Randomisation (week 20) to week 68
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 491 | 233
Ratio of Calcitonin | 1.00 (24.8) | 0.95 (25.5)

ADVERSE EVENTS:
Time Frame: week 0 to week 75 Results are based on the SAS which included all participants who received at least one dose of semaglutide or placebo.
Description: All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment and no later than the date of last dose + 7 weeks.
Groups:
- Semaglutide: Run-in Period: Participants were to receive once-weekly s.c injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL in run-in period (week 0 to week 20) with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached.
- Semaglutide 2.4: Treatment Period: Participants were to receive once-weekly s.c injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL in 20 week run-in period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. The participants with target dose reached were randomised in 2:1 at week 20. Thus, out of 803, 535 participants were continued to receive once weekly semaglutide s.c 2.4 mg until week 68.
- Placebo: Treatment Period: Participants were to receive once-weekly s.c injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL in 20 week run-in period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. The participants with target dose reached were randomised in 2:1 at week 20. Thus, out of 803, 268 participants were switched to receive once weekly placebo until week 68.
Arm/Group | Semaglutide: Run-in Period | Semaglutide 2.4: Treatment Period | Placebo: Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/902 | 1/535 | 1/268
Serious Adverse Events (participants affected / at risk) | 21/902 | 41/535 | 15/268
Other Adverse Events (participants affected / at risk) | 670/902 | 295/535 | 114/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide: Run-in Period (N=902) | Semaglutide 2.4: Treatment Period (N=535) | Placebo: Treatment Period (N=268)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthroscopic surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Biliary cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 5 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Induced abortion infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Orthognathic surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide: Run-in Period (N=902) | Semaglutide 2.4: Treatment Period (N=535) | Placebo: Treatment Period (N=268)
Abdominal distension (Gastrointestinal disorders) | 50 (53) | 8 (10) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 67 (82) | 34 (45) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 49 (64) | 20 (22) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (23) | 25 (28) | 14 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (28) | 28 (32) | 18 (19)
Constipation (Gastrointestinal disorders) | 200 (232) | 62 (75) | 16 (18)
Decreased appetite (Metabolism and nutrition disorders) | 102 (115) | 7 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 212 (309) | 77 (114) | 19 (26)
Dyspepsia (Gastrointestinal disorders) | 103 (127) | 9 (9) | 2 (2)
Eructation (Gastrointestinal disorders) | 71 (88) | 14 (15) | 1 (1)
Fatigue (General disorders) | 67 (69) | 26 (29) | 6 (6)
Flatulence (Gastrointestinal disorders) | 50 (73) | 14 (44) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 58 (60) | 5 (6) | 1 (1)
Headache (Nervous system disorders) | 96 (119) | 41 (48) | 10 (10)
Influenza (Infections and infestations) | 28 (28) | 39 (45) | 19 (23)
Nasopharyngitis (Infections and infestations) | 92 (102) | 58 (77) | 39 (54)
Nausea (Gastrointestinal disorders) | 422 (629) | 75 (104) | 13 (13)
Vomiting (Gastrointestinal disorders) | 140 (239) | 54 (87) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03548987/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03548987/SAP_001.pdf